CLINICAL TRIAL: NCT01459575
Title: Unboosted Atazanavir as Initial ART Therapy in China
Status: Completed | Type: Observational
Sponsor: National Center for AIDS/STD Control and Prevention, China CDC (Other Government)
Collaborators: BMS company (Unknown)
Responsible Party: Principal Investigator, NCAIDS, National Center for AIDS/STD Control and Prevention, National Center for AIDS/STD Control and Prevention, China CDC
Other Study IDs: ATV 2005
Record Dates: First submitted 2011-10-24; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Antiretroviral Therapy
Keywords: Acquired Immunodeficiency Syndrome; antiretroviral therapy; China
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an open-label, Pilot study.The study hypothesis is that the feasibility and efficacy of a non-boosted ATV based HAART will be well as the first line treatment in a Chinese resource-limited setting.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* The subject should have established HIV infection more than 6 month.
* Qualifying plasma HIV RNA ≥ 2,000 c/mL and a CD4 cell count within 100 - 350 cells/mm3
* ≥16 years of age
* Both females of child-bearing potential and males must utilize effective barrier contraception - other contraception in addition to barrier methods are permitted
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

* Patients who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the study.
* Presence of a newly diagnosed HIV-related opportunistic infection or any medical condition requiring acute therapy at the time of enrollment.
* History of hemophilia
* Proven or suspected acute hepatitis in the 30 days prior to study entry. Subjects with chronic hepatitis are eligible provided that their liver function enzymes are < 3 times the upper limit of normal.
* Presence of cardiomyopathy.
* A history of arrhythmia or clinical symptoms potentially related to heart block or second / third degree heart block.
* Inability to tolerate oral medication
* Presence of a newly diagnosed HIV-related opportunistic infection or any medical condition requiring acute therapy at the time of enrollment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ART-naïve patients, established HIV infection > 6 months with CD4 count of 100~350 cell/mm3
Sampling Method: Non-Probability Sample
Dates: Start 2005-07; Primary Completion 2005-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fujie Zhang, MD, Principal Investigator — National Center for AIDS/STD control and prevention
Locations (1):
- Yan Zhao, Beijing, China